CLINICAL TRIAL: NCT05922423
Title: Exploration of Management Model and Intervention Research on Fear of Cancer Recurrence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NFEC-2023-008
Record Dates: First submitted 2023-05-24; First posted 2023-06-28 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Cancer Patients
Keywords: Mindfulness-Based Stress Reduction; fear of cancer recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR (Experimental): Week 1: Introduce mindfulness theory knowledge to participants and guide them to engage in mindfulness breathing training; Week 2: Sitting meditation, explaining the essence of meditation and practicing with music; Week 3: Explain the connotation of walking meditation, inform the participants of precautions, and guide them to practice; Week 4: Explain the connotation and requirements of body scanning, guide participants in practice; Week 5: Introduce the connotation of hatha yoga and guide participants to practice; Week 6: Explain the meaning of mindfulness sounds and thoughts, guide participants to practice; Week 7: Explain the characteristics of non selective perception, combined with music practice; Week 8: Emphasize mindfulness to promote health, encourage participants to practice internalization, and develop into their own patterns.
  Interventions: Behavioral: MBSR
- health education (Placebo Comparator): For cancer patients who have entered the comfort group, automatic tweets and health knowledge related to science popularization will be provided knowledge
  Interventions: Behavioral: health education

INTERVENTIONS:
Behavioral: MBSR — Week 1: Introduce mindfulness theory knowledge to participants and guide them to engage in mindfulness breathing training; Week 2: Sitting meditation, explaining the essence of meditation and practicing with music; Week 3: Explain the connotation of walking meditation, inform the participants of precautions, and guide them to practice; Week 4: Explain the connotation and requirements of body scanning, guide participants in practice; Week 5: Introduce the connotation of hatha yoga and guide participants to practice; Week 6: Explain the meaning of mindfulness sounds and thoughts, guide participants to practice; Week 7: Explain the characteristics of non selective perception, combined with music practice; Week 8: Emphasize mindfulness to promote health, encourage participants to practice internalization, and develop into their own patterns.
  Arms: MBSR
Behavioral: health education — For cancer patients who have entered the comfort group, automatic tweets and health knowledge related to science popularization will be provided knowledge
  Arms: health education

SUMMARY:
1. Through cross-sectional investigation and research, construct an fear of cancer recurrence warning model to identify and screen high fear of cancer recurrencecancer populations, in order to identify predictive factors for high fear of cancer recurrence, study how cancer patients develop susceptibility to fear of cancer recurrence during the diagnosis and treatment process, including which participating factors, explore the development trajectory of fear of cancer recurrence, and effectively prevent the occurrence of high-level fear of cancer recurrence.
2. Through randomized controlled trials, conduct a study on mindfulness and stress reduction psychosocial intervention for high-level fear of cancer recurrence patients, verify the effectiveness of psychosocial intervention measures targeting domestic cancer populations, and improve standardized intervention methods, intervention time, and treatment content.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years old
* Consistent with pathological diagnosis of cancer
* Able to understand and comply with research protocols
* Written informed consent can be provided
* Own and know how to use smart ·terminals (such as smartphones, tablets, computers, etc.)

Exclusion Criteria:

* Patients with mental illness and consciousness disorders;
* Patients with cancer metastasis or recurrence
* End of life treatment for patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fear of cancer recurrence | Baseline
  subjects' fear of cancer recurrence indicators at baseline
Fear of cancer recurrence | At the end of the 8-week intervention
  Change in fear of cancer recurrence score compared to baseline at 8 weeks.
Fear of cancer recurrence | 1 mouth
  Fear of cancer recurrence after one month of intervention
Fear of cancer recurrence | 3 months
  Fear of cancer recurrence after three months of intervention

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT05922423/ICF_000.pdf